CLINICAL TRIAL: NCT01120977
Title: Reference Values for Body Composition Parameters and IGF-I in the Adult NordiNet® International Outcome Study
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 25274
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample to measure "Insulin like growth factor-1" (IGF-1)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Male
- Female

SUMMARY:
The treatment of Growth Hormone deficiency (GHD) patients with GH, often induce fluid retention; this effect is dose dependent and temporary. The symptoms are swelling of soft tissue and joint stiffness. The objective of this study is to create bioelectric impedance/arm muscle area (BIA/AMA) reference data, as a measurement of hydration status, of healthy persons of both genders in the age 20-70 years.

DETAILED DESCRIPTION:
The treatment of Growth Hormone deficiency (GHD) patients with GH, has since 1994 been approved in several countries. The approval is based on studies that show positive effect on body composition, physiology, lipid profile, bone density and life quality. One often observed side effect is fluid retention; this effect is dose dependent and temporary. The symptoms are swelling of soft tissue and joint stiffness.

By comparing the body bioelectric impedance (BIA) with an Arm Muscle Area (AMA) measurement, it is possible to determine the hydrations status of a person. This measurement is a simple and non invasive method to evaluate the GH dosages applied in the treatment of GHD persons.

The objective of this study is to create BIA/AMA reference data of healthy persons of both genders in the age 20-70 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons,
* Age 20- 70 years.

Exclusion Criteria:

* Cardiac implanter (pacemaker),
* Heart insufficiency, chronic venuos insufficiency,
* Use of diuretics, desmopressin, neuroleptica, antidepressants, corticosteroids, fludrocotidon,
* Obesity (BMI > 30),
* Knowledge of changes in electrolyte or water homeostasis.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects are healthy persons in the age 20-70 years, both males and females will be recruited from the city Aarhus in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens O Jørgnsen, Professor, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus university hospital NBG, Aarhus, Denmark